CLINICAL TRIAL: NCT00630305
Title: Evaluation of the Short-Term Corneal Endothelial Response to Wear of Toric Soft Contact Lenses in Asian Eyes
Brief Title: Endothelial Bleb Response With Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0726; JJO0717
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Ametropia
Keywords: toric; endothelial bleb
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Session A (Other): Subjects were first randomized to a session and then randomized to receive one of four lens sequences for that session. Each subject participated in all four sessions. Session A only contains senofilcon A toric and alphafilcon A toric lenses.
  Interventions: Device: alphafilcon A toric; Device: senofilcon A toric
- Session B (Other): Subjects were first randomized to a session and then randomized to receive one of four lens sequences for that session. Each subject participated in all four sessions. Session B only contains senofilcon A toric and alphafilcon A toric lenses.
  Interventions: Device: alphafilcon A toric; Device: senofilcon A toric
- Session C (Other): Subjects were first randomized to a session and then randomized to receive one of four lens sequences for that session. Each subject participated in all four sessions. Session C only contains senofilcon A toric and lotrafilcon B toric lenses.
  Interventions: Device: lotrafilcon B toric; Device: senofilcon A toric
- Session D (Other): Subjects were first randomized to a session and then randomized to receive one of four lens sequences for that session. Each subject participated in all four sessions. Session D only contains senofilcon A toric and lotrafilcon B toric lenses.
  Interventions: Device: lotrafilcon B toric; Device: senofilcon A toric

INTERVENTIONS:
Device: alphafilcon A toric — Subjects that were randomized to receive alphafilcon A toric during one of the four sessions (Sessions A, B, C and D).
  Arms: Session A; Session B
Device: lotrafilcon B toric — Subjects that were randomized to receive lotrafilcon B toric during one of the four sessions (Sessions A, B, C and D).
  Arms: Session C; Session D
Device: senofilcon A toric — Subjects that were randomized to receive senofilcon A toric during one of the four sessions (Sessions A, B, C and D).

SUMMARY:
Evaluate the short-term corneal response of oxygen deprivation when using toric contact lenses. The response will be noted by endothelial bleb formation in both open eye and closed eye state.

DETAILED DESCRIPTION:
Interested subjects who meet the entry criteria for the study will be scheduled for four sessions of approximately 30 minutes duration each. Informed consent obtained. Baseline measurements of visual acuity and corneal and conjunctival physiology will be recorded. An examination of the endothelium of the corneas will be conducted using the specular microscope, readings obtained at 5 locations on each cornea: one in the centre and one in each of the superior, inferior, nasal and temporal peripheral regions, approximately 2mm from the limbal margin. The assigned lenses will be inserted according to a fixed-allocation randomization schedule, where each session follows an optimized 2- period simultaneous crossover design, which specifies lenses to be used in each of the four sessions. Lenses will be worn for 20 minutes and then removed. Endothelial specular microscopy will be conducted at 20 minutes with the lenses on. A final evaluation of corneal and conjunctival physiology will be performed prior to subject clearance from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Successful soft contact lens wear in daily mode for a minimum of 1 month prior to start of the study without experiencing difficulties or contact lens related complications.
2. At least 18 years of age and mentally competent to sign an informed consent form.
3. Healthy eyes and no use of ocular medication.
4. Similarity of optical parameters between eyes.
5. Physical appearance typical of Asian eyes

Exclusion Criteria:

1. A medical or ocular condition that may influence the outcome of this trial.
2. Current use of ocular/systemic medication that may influence the outcome of this trial.
3. Failure to wear soft lenses for 2 weeks prior to the start of the study.
4. Current enrolment or participation in another clinical study.
5. Current state of pregnancy or breastfeeding
6. Anisometropia greater than 1.00D (equivalent sphere).
7. Unequal acuities between eyes (greater than 1 line)
8. Unequal corneal curvatures (>1.00D)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel A Brennan, McOptom PhD, Principal Investigator — Brennan Consultants
Locations (1):
- Brennan Consultants 110 Auburn Rd, Auburn Village, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 37 subjects enrolled, with two being discontinued. Thirty-five (35) subjects were recruited to a single site, where eligibility was confirmed and informed consent discussed and when appropriate signed.
Pre-assignment Details: Subjects were randomized to go to all four sessions (A, B, C and D) in a random order. Once in a session subjects were further randomized to one of four contralteral lens sequences (right eye / left eye).
Groups:
- Overall: subjects were randomized to a session (A, B, C and D) and then to one of four lens sequences. Each subject participated in every session.
Period: Overall Study
Arm/Group | Overall
Started | 37
Completed | 35
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Inability to insert contact lens | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and randomized to a trial arm.
Groups:
- All Subjects: All subjects who were enrolled, randomized, and assigned to a study arm.
Arm/Group | All Subjects
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (7.7)
Gender [Count of Participants; unit: Participants]
  Female | 25
  Male | 12
Region of Enrollment [Number; unit: participants]
  Australia | 37

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Bleb Areas on Cornea: Session A- Open Eye
Description: Mean area of endothelial blebs in the following corneal locations: Central, Nasal, Temporal, Inferior, Superior. A masked observer performed the analysis by subjectively selecting a region in a given image that provided an optimal balance of maximum area and clarity of cell outlines. Blebs were then outlined manually and the software calculated the area of blebs. The different sessions are reported showing results for each lens according to the lens worn in the contralateral (contra) eye.Open eye sessions simulated the subjects normal ocular behavior during waking hours; closed eye sessions simulated ocular activity during duration of closed eye activity, such as sleeping. Results are reported as the mean percent difference between the stated test (senofilcon A) and the control lens (alphafilcon A, lotrafilcon B), after 20 minutes of wear, for each testing scenario.
Time Frame: 20 minutes post-lens insertion
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation. The analysis was conducted on subject eyes.
Measure: Mean (Standard Deviation); unit: Percent Difference of Bleb Area
Units Other Than Participants: Subjects Eyes
Groups:
- Sequence 1: Subjects that first received senofilcon A in their right eye and then received alphafilcon A in their left eye.
- Sequence 2: Subjects that first recieved alphafilcon A in their right eye and then received senofilcon A in their left eye.
- Sequence 3: Subjects that first received senofilcon A in their right eye and then received senofilcon A in their left eye.
- Sequence 4: Subjects that first received alphafilcon A in their right eye and then received alphafilcon A in their left eye.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Subjects Eyes) | 68 | 68 | 68 | 68
Percent Difference of Bleb Area
  Central | 0.1 (0.1) | 2.0 (0.1) | 0.2 (0.1) | 2.1 (0.7)
  Inferior | 0.0 (0.0) | 0.8 (0.3) | 0.1 (0.0) | 2.3 (1.0)
  Nasal | 0.0 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.7 (0.4)
  Superior | 0.2 (0.1) | 0.0 (0.0) | 0.0 (0.0) | 0.3 (0.1)
  Temporal | 0.0 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.4 (0.2)

2. Primary Outcome: Endothelial Bleb Areas on Cornea: Session B- Closed Eye
Description: as for outcome 1
Time Frame: 20 minutes post-lens insertion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Difference of Bleb Area
Units Other Than Participants: Subject Eyes
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Subject Eyes) | 68 | 68 | 68 | 68
Percent Difference of Bleb Area
  Central | 2.0 (0.9) | 5.9 (2.5) | 4.0 (0.9) | 0.9 (0.5)
  Inferior | 0.5 (0.3) | 3.9 (2.2) | 2.5 (0.5) | 0.9 (0.3)
  Nasal | 0.5 (0.3) | 0.9 (0.1) | 1.0 (0.3) | 0.1 (0.1)
  Superior | 0.1 (0.0) | 0.2 (0.) | 10.3 (0.1) | 0.3 (0.1)
  Temporal | 0.2 (0.1) | 0.5 (0.2) | 0.5 (0.2) | 0.3 (0.1)

3. Primary Outcome: Endothelial Bleb Areas on Cornea: Session C- Open Eye
Description: as for outcome 1
Time Frame: 20 minutes post-lens insertion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Difference of Bleb Area
Units Other Than Participants: Subject Eyes
Groups:
- Sequence 1: Subjects that first received senofilcon A in their right eye and then received lotrafilcon B in their left eye.
- Sequence 2: Subjects that first recieved lotrafilcon B in their right eye and then received senofilcon A in their left eye.
- Sequence 4: Subjects that first received lotrafilcon B in their right eye and then received lotrafilcon B in their left eye.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Subject Eyes) | 68 | 68 | 68 | 68
Percent Difference of Bleb Area
  Central | 0.2 (0.1) | 0.4 (0.3) | 0.2 (0.1) | 0.2 (0.1)
  Inferior | 0.1 (0.0) | 0.1 (0.1) | 0.1 (0.0) | 0.1 (0.0)
  Nasal | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.2 (0.1)
  Superior | 0.1 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.4 (0.1)
  Temporal | 0.0 (0.0) | 0.1 (0.0) | 0.0 (0.0) | 0.1 (0.0)

4. Primary Outcome: Endothelial Bleb Areas on Cornea: Session D- Closed Eye
Description: as for outcome 1
Time Frame: 20 minutes post-lens insertion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Difference of Bleb Area
Units Other Than Participants: Subject Eyes
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (Subject Eyes) | 68 | 68 | 68 | 68
Percent Difference of Bleb Area
  Central | 1.7 (0.6) | 1.6 (0.6) | 0.5 (0.2) | 3.5 (2.0)
  Inferior | 0.8 (0.3) | 1.7 (1.0) | 0.3 (0.1) | 1.4 (0.7)
  Nasal | 0.2 (0.1) | 0.8 (0.4) | 0.1 (0.1) | 0.7 (0.3)
  Superior | 0.2 (0.1) | 0.1 (0.1) | 0.3 (0.2) | 0.1 (0.1)
  Temporal | 0.1 (0.1) | 0.2 (0.1) | 0.1 (0.0) | 0.3 (0.1)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study.
Groups:
- Session A: Open eye session, this session includes the following sequences only:
  1. senofilcon A / alphafilcon A
  2. alphafilcon A / senofilcon A
  3. senofilcon A / senofilcon A
  4. alphafilcon A / alphafilcon A
- Session B: Closed eye session, this session includes the following sequences only:
  1. senofilcon A/ alphafilcon A
  2. alphafilcon A/ senofilcon A
  3. senofilcon A/ senofilcon A
  4. alphafilcon A/ alphafilcon A
- Session C: Open eye session, this session includes the following sequences only:
  1. senofilcon A/ lotrafilcon B
  2. lotrafilcon B / senofilcon A
  3. senofilcon A/ senofilcon A
  4. lotrafilcon B / lotrafilcon B
- Session D: Closed eye session, this session includes the following sequences only:
  1. senofilcon A/ lotrafilcon B
  2. lotrafilcon B / senofilcon A
  3. senofilcon A/ senofilcon A
  4. lotrafilcon B / lotrafilcon B
Arm/Group | Session A | Session B | Session C | Session D
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other